CLINICAL TRIAL: NCT01718184
Title: Piggyback Sulcoflex Toric IOL for Correcting Refractive Error Following Corneal Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Collaborators: Einat Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RabinMC Sulcoflex Toric IOL
Record Dates: First submitted 2012-10-29; First posted 2012-10-31 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-07

CONDITIONS: Refractive Error; Corneal Implantation; Intraocular Lens Implantation
Keywords: sulcoflex; toric; corneal implantation
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sulcoflex (Experimental): Sulcoflex intraocular lens implantation
  Interventions: Procedure: toric intraocular lens implantation; Procedure: Sulcoflex intraocular lens implantation

INTERVENTIONS:
Procedure: toric intraocular lens implantation — piggyback Sulcolflex toric intraocular lens implantation
Procedure: Sulcoflex intraocular lens implantation

SUMMARY:
A prospective study to evaluate the safety and efficacy of a piggyback sulcoflex toric intraocular lens in pseudophakic patients for correcting refractive errors following corneal transplantation

ELIGIBILITY:
Inclusion Criteria:

* after corneal transplantation with refractive errors
* after cataract removal and intraocular lens implantation

Exclusion Criteria:

* other ophthalmologic disorders limiting vision including glaucoma, AMD, profound amblyopia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-04 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Best corrected and uncorrected visual acuity | 3 month
  Best corrected and uncorrected visual acuity following the IOL implantation

SECONDARY OUTCOMES:
Ocular complications | 3 months
  pigmentary dispersion, iris bulging, inter lenticular opacifications, lens decentration

OTHER OUTCOMES:
Refractive outcomes | 3 months
  refractive outcomes following surgical intervention

CONTACTS AND LOCATIONS:
Overall Officials: Irit Bahar, MD, Principal Investigator — Rabim Medical Center, Israel
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

REFERENCES:
- [Background] Leaming DV. Practice styles and preferences of ASCRS members--2003 survey. J Cataract Refract Surg. 2004 Apr;30(4):892-900. doi: 10.1016/j.jcrs.2004.02.064. PMID 15093657
- [Background] Mamalis N, Brubaker J, Davis D, Espandar L, Werner L. Complications of foldable intraocular lenses requiring explantation or secondary intervention--2007 survey update. J Cataract Refract Surg. 2008 Sep;34(9):1584-91. doi: 10.1016/j.jcrs.2008.05.046. PMID 18721724
- [Background] Paul RA, Chew HF, Singal N, Rootman DS, Slomovic AR. Piggyback intraocular lens implantation to correct myopic pseudophakic refractive error after penetrating keratoplasty. J Cataract Refract Surg. 2004 Apr;30(4):821-5. doi: 10.1016/j.jcrs.2003.08.008. PMID 15093644
- [Background] Gayton JL, Sanders VN. Implanting two posterior chamber intraocular lenses in a case of microphthalmos. J Cataract Refract Surg. 1993 Nov;19(6):776-7. doi: 10.1016/s0886-3350(13)80349-5. PMID 8271176
- [Background] Gayton JL. Secondary implantation of a double intraocular lens after penetrating keratoplasty. J Cataract Refract Surg. 1998 Feb;24(2):281-2. doi: 10.1016/s0886-3350(98)80212-5. PMID 9530606
- [Background] Gayton JL, Sanders V, Van der Karr M, Raanan MG. Piggybacking intraocular implants to correct pseudophakic refractive error. Ophthalmology. 1999 Jan;106(1):56-9. doi: 10.1016/S0161-6420(99)90005-2. PMID 9917781
- [Background] Habot-Wilner Z, Sachs D, Cahane M, Alhalel A, Desatnik H, Schwalb E, Barequet IS. Refractive results with secondary piggyback implantation to correct pseudophakic refractive errors. J Cataract Refract Surg. 2005 Nov;31(11):2101-3. doi: 10.1016/j.jcrs.2005.05.023. PMID 16412922
- [Background] Werner L, Shugar JK, Apple DJ, Pandey SK, Escobar-Gomez M, Visessook N, Evans BB. Opacification of piggyback IOLs associated with an amorphous material attached to interlenticular surfaces. J Cataract Refract Surg. 2000 Nov;26(11):1612-9. doi: 10.1016/s0886-3350(00)00485-5. PMID 11084268
- [Background] Werner L, Apple DJ, Pandey SK, Solomon KD, Snyder ME, Brint SF, Gayton JL, Shugar JK, Trivedi RH, Izak AM. Analysis of elements of interlenticular opacification. Am J Ophthalmol. 2002 Mar;133(3):320-6. doi: 10.1016/s0002-9394(01)01405-2. PMID 11860967
- [Background] Baumeister M, Kohnen T. Scheimpflug measurement of intraocular lens position after piggyback implantation of foldable intraocular lenses in eyes with high hyperopia. J Cataract Refract Surg. 2006 Dec;32(12):2098-104. doi: 10.1016/j.jcrs.2006.08.033. PMID 17137990
- [Background] Chang SH, Lim G. Secondary pigmentary glaucoma associated with piggyback intraocular lens implantation. J Cataract Refract Surg. 2004 Oct;30(10):2219-22. doi: 10.1016/j.jcrs.2004.03.034. PMID 15474839
- [Background] Chang WH, Werner L, Fry LL, Johnson JT, Kamae K, Mamalis N. Pigmentary dispersion syndrome with a secondary piggyback 3-piece hydrophobic acrylic lens. Case report with clinicopathological correlation. J Cataract Refract Surg. 2007 Jun;33(6):1106-9. doi: 10.1016/j.jcrs.2007.01.044. PMID 17531710
- [Background] Iwase T, Tanaka N. Elevated intraocular pressure in secondary piggyback intraocular lens implantation. J Cataract Refract Surg. 2005 Sep;31(9):1821-3. doi: 10.1016/j.jcrs.2005.06.034. PMID 16246790
- [Background] Durak I, Ferliel ST, Soylev M, Saatci O. Pre-Descemet's membrane hemorrhage after secondary intraocular lens implantation. J Cataract Refract Surg. 1999 Nov;25(11):1554-6. doi: 10.1016/s0886-3350(99)00249-7. PMID 10569176
- [Background] Kahraman G, Amon M. New supplementary intraocular lens for refractive enhancement in pseudophakic patients. J Cataract Refract Surg. 2010 Jul;36(7):1090-4. doi: 10.1016/j.jcrs.2009.12.045. PMID 20610084
- [Background] Khan MI, Muhtaseb M. Performance of the Sulcoflex piggyback intraocular lens in pseudophakic patients. J Refract Surg. 2011 Sep;27(9):693-6. doi: 10.3928/1081597X-20110512-01. Epub 2011 May 20. PMID 21598871
- [Background] McIntyre JS, Werner L, Fuller SR, Kavoussi SC, Hill M, Mamalis N. Assessment of a single-piece hydrophilic acrylic IOL for piggyback sulcus fixation in pseudophakic cadaver eyes. J Cataract Refract Surg. 2012 Jan;38(1):155-62. doi: 10.1016/j.jcrs.2011.06.035. Epub 2011 Nov 4. PMID 22055074